CLINICAL TRIAL: NCT04742270
Title: Feasibility of Implementing SIMEOX® Using Tele-physiotherapy and Evaluation of Compliance With SIMEOX® at Home for Bronchial Drainage in Patients With Bronchiectasis Other Than Cystic Fibrosis and Who Have Difficulties in Accessing Regular Respiratory Physiotherapy Sessions.
Brief Title: Home Airway Clearance in Patients With Bronchiectasis (Home-Care Bronchiectasis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Collaborators: Icadom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-03
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Bronchiectasis Adult
Keywords: Airway Clearance; Bronchiectasis; Respiratory Physiotherapy Telecare
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: There is no comparison procedure included in this feasibility trial. Patients will be their own control.
Masking Description: Non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIMEOX+ respiratory physiotherapy telecare (Experimental): Use the device for 3 months in addition to usual care
  Interventions: Device: SIMEOX+ respiratory physiotherapy telecare

INTERVENTIONS:
Device: SIMEOX+ respiratory physiotherapy telecare — Every 10 days, the patient's expert physiotherapist will contact the patient by video-transmission or telephone call for motivational reinforcement and technical support in the use of the device.
  During these phone calls, a quick 3-question questionnaire will be administered to the patient to monitor events of hemoptysis, chest pain and clinical symptoms of gastroesophageal reflux disease: pyrosis.If patients report this type of event, the physiotherapist will inform the patient's physician for management at his/her discretion.
  The expert physiotherapist will also conduct this sessions in order to increase the patient's motivation and compliance to the device. In order to do this, he will identify (in collaboration with the patient), the patient's difficulties and obstacles and he will try to find solutions with him.

SUMMARY:
Bronchiectasis is a chronic multiple etiologies pulmonary disease characterized by permanent dilatation of the caliber of the bronchial tree territory with an alteration of mucociliary clearance. This alteration causes mucus retention and leads to infections and chronic bronchial inflammation. Respiratory physiotherapy is one of the cornerstones of the management of these patients, particularly to facilitate bronchial drainage. In patients with abundant bronchial secretions, it is recommended to carry out airway clearance sessions daily or several times a day, which represents a very significant burden of care. Moreover, access to respiratory physiotherapy care isn't always easy for patients due to geographical, time, or professional availability limitations. In addition, few professionals are trained in France for this specific care dedicated to chronic lung disease. Finally with this kind of remote formation and follow up, it may be more suitable for this at-risk patient population in the context of the COVID-19 pandemic situation (limitation of physical contact).

SIMEOX® (Physio-Assist, Aix en Provence, France) is an innovative medical device (CE medical mark) for bronchial tree drainage. The use of this device in autonomy by the patient requires however a specific initial training of a few sessions (3-5 sessions). Tele-physiotherapy could allow remote training of patients in the use of SIMEOX®. This SIMEOX® device used autonomously at home, could provide patients with a practical and efficient bronchial clearance technique.

The overall objective of this pilot study is to evaluate the use of SIMEOX® at home after education in its use by telecare for bronchial drainage in patients with bronchiectasis (non-cystic Fibrosis Bronchiectasis) and who have difficulty accessing usual respiratory physiotherapy sessions.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic multiple etiologies pulmonary disease characterized by permanent and abnormal dilatation of the caliber of a territory of the bronchial tree with an alteration of mucociliary clearance. Patients with bronchiectasis have chronic cough and sputum production. Bacterial infections develop in them, leading to loss of lung function. Bronchiectasis affects patients of all ages and sexes, but the prevalence is higher in older women. It is often a complication of a previous lung infection or injury or is due to underlying systemic diseases. The treatment of bronchiectasis is multimodal and non-specific, including anti-inflammatory agents, bronchodilation, and depending on the clinical picture, bronchodilators, and inhaled antibiotics.

Respiratory physiotherapy is one of the cornerstones to facilitate bronchial drainage. In patients with abundant bronchial secretions, it is recommended that bronchial drainage sessions be performed daily or several times a day. These bronchial drainage sessions, whether performed with a physiotherapist or independently, represent a very significant burden of care with limited compliance. Moreover, access to respiratory physiotherapy care is not always easy for patients due to geographical, time or professional availability limitations. Telehealth is recommended to improve the access to care and the quality of care. The Article 53 of French Law No. 2019-774 of July 24, 2019, relating to the organization and transformation of the healthcare system, provides for telecare. In the context of respiratory physiotherapy, this is a session carried out remotely by the physiotherapist, by videotransmission. In the context of the COVID-19 health crisis, this telecare was regulated by the decree of May 11, 2020. The rehabilitation of respiratory diseases (excluding emergencies) was envisaged in this decree. Practical experiences of telecare in respiratory physiotherapy have emerged during this health crisis and have created an opportunity to facilitate access to care for patients.

The general principle expected from bronchial clearance techniques is to modify the viscoelastic properties of secretions and facilitate their elimination; these techniques can be applied simply with the spontaneous breathing of the patient by modifying the respiratory flow and/or the amplitude of ventilation or they can be applied with instrumental aids. SIMEOX® (Physio-Assist, Aix en Provence, France) is an innovative medical device (CE medical mark) for drainage of the bronchial tree: by means of a mouthpiece connected to SIMEOX® a succession of very short air negative pressure are generated in a non-invasive way that disseminate in the bronchial tree a pneumatic vibratory signal that modifies the rheological properties of the mucus, facilitates the mobilization of secretions and assists their transport to the upper airways. The SIMEOX® device was tested in patients with bronchiectasis during respiratory exacerbation during a 7-day hospital stay; patients reported good tolerance of the device; respiratory function and exercise tolerance parameters were improve. However, the patient's autonomous use of this device requires specific training of a few sessions (3 to 5 sessions).

RESEARCH HYPOTHESES Tele-physiotherapy could allow remote training of patients in the use of SIMEOX®. Once trained in its use, patients who have difficulty accessing standard respiratory physiotherapy sessions could be provided with a practical and effective bronchial clearance technique that can be used independently at home.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of bronchiectasis confirmed by HR CT scan, regardless of etiology except cystic fibrosis and with estimated bronchorrhea >10mL/d.
* Disease stability, defined as a delay of at least 4 weeks since the end of an exacerbation (end of antibiotic therapy or judged as resolved by the investigator).
* Age > 18 years old
* Patient does not have access to a physiotherapist or does not usually go to a physiotherapy office (<1/week on average)

Exclusion Criteria:

* Pneumothorax or severe hemoptysis (more than 30 ml per 24 hours) within 6 weeks before inclusion,
* Patient on transplant list
* Any contraindication to an instrumental bronchial clearance technique (at the discretion of the investigator)
* Patient not available or wishing to change of region within 3 months of inclusion
* Patient is currently participating or has participated within one month prior to inclusion in another clinical intervention research study that may impact the study, the impact of which is at the discretion of the investigator.
* Persons referred to in articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: pregnant woman (verified by the dosage of β-HCG for any woman wishing to participate in the protocol and of childbearing age < 60 years), parturient, breastfeeding mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Compliance | 3 months after inclusion
  The compliance with the SIMEOX® device at home is assessed by the change in the percentage of patient with an average of at least 3 sessions/week between D15 and 3 months (self-reported compliance by the patient on a diary)

SECONDARY OUTCOMES:
Compliance reliability | 3 months after inclusion
  Comparison of self-reported patient compliance to compliance reported on the "Simeox web application" web platform is assessed by the variation between the total number of sessions self-reported by the patient via a diary and the number of sessions found on the secure web platform "Simeox web application" between D15 and 3 months
Device use | 3 months after inclusion
  The evolution of the use of the device (number of sessions self-reported by the patient) between D15 and 3 months will be described per week for all patients
Device satisfaction | 3 months after inclusion
  Patient satisfaction with the SIMEOX device will be estimated using a visual analog scale from 0 for the worst satisfaction to 10 for the best satisfaction.
General compliance | At inclusion
  Overall therapeutic adherence will be estimated by the BMQ questionnaire (Beliefs about Medecines Questionnaire) from 5 for the worst general compliance to 25 for the best general compliance.
Link between compliance to treatment and Physical activity | At inclusion and 3 months after
  The link between treatment compliance and physical activity will be assessed by the IPAQ questionnaire (International Physical Activity Questionnaire). This questionnaire provides separate scores on sedentary, walking, moderate-intensity, and vigorous-intensity activity.
Poor compliance factors | At inclusion
  To determine the factors associated with poor (self-reported) compliance with the SIMEOX® device.
  Correlations between insufficient adherence (self-reported; <3 sessions/weeks between D15-D+3 months) to the SIMEOX® device and the following six factors will be sought (age, gender, marital status, socio-professional category, (8 INSEE posts https://www.insee.fr/fr/information/2400059), smoking status, number of drug treatments, severity of bronchiectasis (BSI Score -Bronchiectasia Severity Index), co-morbidities.
Sputum collection feasability | 3 months after inclusion
  To evaluate the feasibility of a weekly collection by the patient of the quantity of bronchial secretions after a bronchial clearance session with SIMEOX®.
  The feasibility of a weekly collection by the patient will be estimated by the frequency and weight of secretions reported on the patient's diary.
Quality of session | 3 months after inclusion
  To assess the link between the quality of the session found on the web platform and the efficiency of bronchial clearance estimated by the frequency and weight of secretions reported on the patient's diary.
Tele-physiotherapy feasability | 3 months after inclusion
  To evaluate the feasibility of one call every 10 days (reported by the patient in his or her diary) for therapeutic motivational reinforcement.
Specific quality of life | At inclusion and 3 months after
  To evaluate the effect of SIMEOX®+ tele-physiotherapy on the specific quality of life of bronchiectasis after 3 months of home treatment.
  The variation in quality of life will be measured by the change of the Qol-B questionnaire's score (total score and respiratory sub-scores, activity, social functioning, vitality, emotional function, constraints related to treatment) between inclusion and 3 months after inclusion.
  Score range from 0 to 100, with higher score representing fewer symptoms or better functioning.
Global quality of life | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on the overall quality of life of respiratory diseases after 3 months of home treatment; The change in overall quality of life for respiratory diseases will be measured before and after 3 months of treatment using the Saint Georges Questionnaire (SGQOL).
  Each response to the questionnaire is assigned a unique " value " derived from anterior data. The minimum weight is 0 and the highest is 100. For each component, sum the values assigned to each response. The score is calculated by dividing this sum of the values by the maximum possible score for each component and expressing the result as a percentage.
Cough perception | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on the perception of cough after 3 months of home treatment;The change in cough perception will be measured before and after 3 months of treatment with the Leicester questionnaire.
  It consists of 19 items with a 7 point likert response scale (range from 1 to 7). Each item is developed to assess symptoms during cough and impact of cough on three main domains: physical, psychological and social. Scores are calculated as a mean of each domain and the total score is calculated by adding every domain score.
Bronchial clearance perception | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on the perception of bronchial congestion after 3 months of home treatment;The change in perception of bronchial congestion will be measured before and after 3 months of treatment by the Chronic Airways Assessment Test (CAT) questionnaire.
  Score range from 0 to 40, with higher score representing better health.
Respiratory function :Variation of forced expiratory volume in 1 second (FEV1) | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on respiratory function after 3 months of home treatment on the forced expiratory volume in 1 second (FEV1)
Respiratory function :Pulmonary forced vital capacity (FVC) | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on respiratory function after 3 months of home treatment on relative variation of forced vital capacity in liter
Respiratory function :FEV1/ FVC ratio | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on respiratory function after 3 months of home treatment on relative variation of FEV1/ FVC ratio in %
Respiratory function : Forced Expiratory Flow (FEF) | At inclusion and 3 months after
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on respiratory function after 3 months of home treatment on relative variation of FEF in %
Exacerbation | 3 months after inclusion
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on the number of respiratory exacerbations; Respiratory exacerbations will be documented by the investigating physicians according to the EMBARC consensus definition.
First exacerbation onset | 3 months after inclusion
  Evaluate the effect of SIMEOX®+ tele-physiotherapy on the time to onset of the first respiratory exacerbation.The date of consultation and/or hospitalization attesting to the exacerbation will be documented in the e-CRF to estimate the time to first exacerbation.
Adverse events | 3 months after inclusion
  Adverse events and device causality will be monitored through a questionnaire of 4 items (hemoptysis, chest pain, gastro-esophageal reflux, other) during tele-physiotherapie sessions and eventual event will be collected in the eCRF

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hamidfar, MD, Principal Investigator — Grenoble university affiliated hospital : pneumology department
Locations (3):
- France (3):
  - Grenoble University-Affiliated Hospital : Pneumology department, Grenoble
  - Nice university-affiliated hospital : pneumonoly department, Nice
  - Toulouse University-Affiliated Hospital : Pneumology department, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamidfar R, Murris-Espin M, Mahot M, Abouly R, Gauchez H, Jacques S, Joffray E, Arnol N, Morin L, Leroy S, Borel JC. Feasibility of home initiation of an airway clearance device (SIMEOX) by telecare in people with non-cystic fibrosis bronchiectasis: a pilot study. BMJ Open Respir Res. 2023 Jul;10(1):e001722. doi: 10.1136/bmjresp-2023-001722. PMID 37524523